CLINICAL TRIAL: NCT03650348
Title: A Phase 1b, Open-Label, Dose Escalation Study of PRS-343 in Combination With Atezolizumab in Patients With HER2-Positive Advanced or Metastatic Solid Tumors
Brief Title: PRS-343 in Combination With Atezolizumab in HER2-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRS-343-PCS_08_18
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2-positive Bladder Cancer; HER2-positive Solid Tumor
Keywords: HER2-positive breast cancer; HER2-positive gastric cancer; HER2-positive bladder cancer; Pieris; PRS-343; Anticalin; Bispecific; 4-1BB; CD137; HER2; Atezolizumab
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Drug PRS-343 Combination Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRS-343 in Combination with Atezolizumab (Experimental)
  Interventions: Drug: PRS-343 in Combination with Atezolizumab

INTERVENTIONS:
Drug: PRS-343 in Combination with Atezolizumab — HER2/4-1BB Bispecific

SUMMARY:
A Phase 1b, open-label, dose escalation study of PRS-343 in combination with atezolizumab in patients with HER2-positive advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1b study to determine the MTD and RP2D and to assess the safety and efficacy of PRS-343 administered in combination with atezolizumab, a PD-L1 antibody, in previously treated advanced or metastatic HER-2 positive solid tumors (e.g., bladder, breast and gastrointestinal). The study will include a dose escalation period followed by an expansion period. PRS-343 and atezolizumab will be given intravenously once every three weeks (Q3W).

All available safety data, emerging PK, pharmacodynamic data, and dose limiting toxicities (DLTs) will be considered in guiding the Safety Committee's decisions regarding subsequent doses to be tested during the escalation phase of the study. Once the MTD and RP2D have been established, an expansion cohort will be enrolled.

One treatment cycle is defined as 21 days (3 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to performing any study procedure, including screening procedures.
2. Men and women ≥18 years.
3. Histologically or cytologically confirmed diagnosis of previously treated locally advanced and/or metastatic HER2+ solid tumor malignancy considered likely to respond to a HER2-targeted CD137 agonist (e.g. gastric/gastroesophageal/esophageal, breast, bladder).
4. HER2+ status documented by clinical pathology report.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
6. Estimated life expectancy of at least 3 months.
7. Measurable disease according to RECIST v1.1.
8. Adequate organ function as defined below:
9. Serum AST and ALT ≤ 2.5 X ULN or ≤ 5 X ULN in the presence of liver metastases.
10. Total serum bilirubin ≤ 1.5 X ULN.
11. Serum creatinine ≤ 2 X ULN OR calculated glomerular filtration rate (GFR) by Cockcroft-Gault formula ≥ 30 mL/min.
12. Hemoglobin ≥ 9 g/dL.
13. ANC ≥ 1500/mm3.
14. Platelet count ≥ 75,000/mm3.
15. Left ventricular ejection fraction (LVEF) determined by echocardiogram or multi-gated acquisition scan ≥ 50%.
16. Any prior cumulative doxorubicin dose must be ≤ 360 mg/m2; prior cumulative epirubicin dose must be ≤ 720 mg/m2.
17. Women of childbearing potential must have a negative serum or urine pregnancy test within 96 hours prior to start of study treatment.
18. Women must not be breastfeeding.
19. Women of childbearing potential must agree to follow instruction for method(s) of contraception for the duration of treatment with study drug PRS 343 and atezolizumab plus 5 months post-treatment completion.
20. Males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment plus 90 days post-treatment completion.

Exclusion Criteria:

1. Known uncontrolled central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are clinically stable off steroids for at least 7 days prior to study treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability.
2. History of acute coronary syndromes, including myocardial infarction, coronary artery bypass graft, unstable angina, coronary angioplasty or stenting within past 24 weeks.
3. History of or current Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system (Appendix B).
4. History of ejection fraction drop below the lower limit of normal with trastuzumab and/or pertuzumab.
5. Medical, psychiatric, cognitive or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study.
6. Any severe concurrent disease or condition (includes active infections, cardiac arrhythmia, interstitial lung disease) that in the judgment of the Investigator would make study participation inappropriate for the patient.
7. Previously known infection with human immunodeficiency virus (HIV); or hepatitis B virus (HBV) or hepatitis C virus (HCV) (unless patients are HBV DNA / HCV RNA negative).
8. Any severe infection within 28 days prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia or active tuberculosis.
9. Administration of live, attenuated vaccines within 28 days before Cycle 1 Day 1 or anticipated need of vaccination with live attenuated vaccine during the study.
10. Need for the treatment of bacterial infection with oral or intravenous (IV) antibiotics within 14 days prior to Cycle 1 Day 1.
11. History of infusion reactions to any component/excipient of PRS-343.
12. History of infusion reactions to any component/excipient of atezolizumab.
13. History of severe hypersensitivity reactions to monoclonal antibodies (mAbs).
14. Systemic steroid therapy (>10 mg daily prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment (note: topical, inhaled, nasal and ophthalmic steroids are not prohibited).
15. Autoimmune disease that has required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
16. Prior organ transplantation including allogeneic or autologous stem-cell transplantation.
17. Has not recovered from the adverse effect of previous anticancer treatments to pre-treatment baseline or Grade 1 except for alopecia, anemia (hemoglobin must meet the study inclusion criteria) and peripheral neuropathy (which must have recovered to ≤ Grade 2) nausea and diarrhea if anti-emetic and anti-diarrheal treatment hasn't been exhausted.
18. Concurrent or previous other malignancy within 5 years of study entry with the exception of cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy.
19. Receipt of investigational treatment within 3 weeks of scheduled Cycle 1 Day 1 (C1D1) dosing.
20. Receipt of cytotoxic chemotherapy within 3 weeks (6 weeks for nitrosoureas and mitomycin C) of scheduled C1D1 dosing.
21. Receipt of radiation therapy within 3 weeks of scheduled Day 1 dosing, unless the radiation comprised a limited field to non-visceral structures (e.g., limb bone metastasis).
22. Receipt of treatment with immunotherapy, biological therapies, hormonal therapies within 3 weeks of scheduled C1D1 dosing.
23. Treatment with targeted small molecules within 5 half-lives of scheduled C1D1 dosing.
24. Receipt of trastuzumab or ado-trastuzumab emtansine or any other experimental drug that engages the same epitope as trastuzumab within 4 weeks of scheduled C1D1 dosing.
25. Receipt of atezolizumab or any other experimental drug that engages the same epitope as atezolizumab within 4 weeks of scheduled C1D1 dosing.
26. Concurrent enrollment in another therapeutic clinical trial.
27. Major surgery within 3 weeks of scheduled C1D1 dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs and recommended Phase 2 dose (RP2D) of PRS-343 administered in combination with atezolizumab | Up to 36 months

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST v1.1 | Up to 36 months
Duration of response (DOR) per RECIST v1.1 | Up to 36 months
Rate of complete response (CR) per RECIST v1.1 | Up to 36 months
Incidence and severity of AEs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03, and changes in clinical laboratory parameters | Up to 36 months
Peak Plasma Concentration (Cmax) | Up to 36 months
Area under the plasma concentration versus time curve (AUC) | Up to 36 months
Time to maximum dose concentration (Tmax) | Up to 36 months
Terminal half life (t1/2) | Up to 36 months
Presence and/or concentration of anti-PRS-343 and anti-atezolizumab antibodies (anti-drug antibodies [ADAs]) | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UCLA Health, Santa Monica, California
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided